CLINICAL TRIAL: NCT05688631
Title: Dietary Antioxidant Intake and Thiol Disulfide Homeostasis Relationship in Type 2 Diabetes Mellitus
Brief Title: Dietary Antioxidants and Thiol Disulfide Homeostasis in T2DM
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Rahime Evra KARAKAYA, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYBU-KARAKAYA001
Record Dates: First submitted 2022-12-10; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2; Antioxidative Stress
Keywords: Diabetes mellitus; Dietary antioxidants; Oxidative stress; Thiol disulfide homeostasis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fasting blood samples of each participants were retained in a biorepository to assess native thiol, total thiol, disulfide and ischemia modified albumin until the analysis as described: To prevent the reduction of 5,5'-dithiobis-(2-nitrobenzoic) acid, the unused reducing sodium borohydride was consumed and removed with formaldehyde, and after the reaction with 5,5'-dithiobis-(2-nitrobenzoic) acid, all thiol groups including the reduced and native thiol groups were determined.IMA level measurement was made within 1 hour after the venous blood samples of the individuals were taken. The samples were incubated at room temperature for 30 minutes and then centrifuged at 3500 rpm for 5 minutes. Final samples were transferred to Eppendorf tubes and stored at -80ºC until analysis. The samples were incubated at room temperature for 30 minutes and then centrifuged at 3500 rpm for 5 minutes. Final samples were transferred to Eppendorf tubes and stored at -80ºC until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic participants (case group): Participants diagnosed with type 2 diabetes mellitus
  Interventions: Other: Dietary antioxidant intake
- Healthy participants (control group): Participants not diagnosed with type 2 diabetes mellitus or any other chronic diseases
  Interventions: Other: Dietary antioxidant intake

INTERVENTIONS:
Other: Dietary antioxidant intake — Decreased intake of dietary antioxidant is associated with decreased thiol disulfide homeostasis parameters in diabetic and healthy participants.

SUMMARY:
This observational study was planned to determine the relationship between dietary antioxidant intake and thiol disulfide homeostasis of individuals with type 2 diabetes. One of the current approaches in medical nutrition therapy of diabetes is to increase the consumption of foods with high antioxidant content in order to strengthen antioxidant defense. Increased dietary antioxidant intake may have both protective and therapeutic effects by reducing the risk of diabetes and preventing complications that may occur. It is known that dynamic thiol disulfide balance can be a good indicator of antioxidant defense in individuals with diabetes, and there are limited studies on this subject.

DETAILED DESCRIPTION:
Power analysis was performed to determine the study sample. In order to reveal a moderate to high level effect for each parameter with 80% power and 5% margin of error, it was found appropriate to work with a total of 68 people, 34 of whom were T2DM and 34 of whom were healthy. In order to keep the sample size higher, a total of 87 individuals, including 40 T2DM and 47 healthy individuals, were included in this study. Individuals who agreed to participate in the study gave their informed consent. Anthropometic measurements (body weight and height) were taken by the researcher. BMI values of individuals were calculated with the formula of body weight (kg)/height (m)2 Routine fasting plasma glucose (FPG), hemoglobin A1c (HbA1c), total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, very low-density lipoprotein (VLDL), non-HDL cholesterol, Total/HDL cholesterol ratio, triglyceride (TG), C-reactive protein (CRP) values were analyzed with blood samples taken by the nurse on an 8 hours of fasting in the morning. Dynamic thiol disulfide balance was determined by native thiol, total thiol and disulfide values and oxidized albumin was determined by IMA values. Food consumption records of individuals were taken to determine dietary antioxidant intake and dietary antioxidant capacity. Oxidative balance score was used to evaluate the exposure of individuals to antioxidants and prooxidants. Descriptive statistics for categorical variables are presented as frequency and percentage. The conformity of the numerical variables to the normal distribution was checked using the Shapiro-Wilk Test. The descriptive statistics of numerical variables were given as mean (±) standard deviation for those with normal distribution, and median interquartile range [IQR] values for those without normal distribution. In the comparison of two independent groups; Independent Sample T Test was used if the data provided the assumptions of the parametric tests, the Mann-Whitney U Test was used if the assumptions of the parametric tests were not met, and the Chi-square Test was used for the comparison of two qualitative groups. Examination of the relationships between quantitative variables was determined by the "Pearson Correlation Coefficient" for those with normal distribution and the Spearman Correlation Coefficient for those who did not. In the interpretation of the correlation coefficient, very weak correlation criteria were used if <0.2, weak correlation between 0.2-0.4, moderate correlation between 0.4-0.6, high correlation between 0.6-0.8, and very high correlation if 0.8>. Statistical significance level was considered as α<0.05, α<0.01, α<0.001 in all calculations and interpretations and hypotheses were established as bidirectional. Statistical analysis of the data was performed with SPSS v26 (IBM Inc., Chicago, IL, USA) statistical package program.

ELIGIBILITY:
Inclusion Criteria (for case group):

* Diagnosis with type 2 diabetes mellitus
* Diabetes age for a maximum of 5 years
* Body mass index (BMI)<30 kg/m^2
* Received and applied medical nutrition therapy and metformin therapy

Inclusion Criteria (for control group):

* Body mass index (BMI) <30 kg/m^2

Exclusion Criteria (for case group):

* Receiving insulin therapy
* Developing diabetes-specific complications
* Smoking tobacco
* Consuming alcohol
* Having end-stage chronic renal failure
* Receiving chemotherapy and/or radiotherapy
* Being in menopause, pregnant and/or lactation period
* Using antioxidant vitamin and mineral supplements

Exclusion Criteria (for control group):

* Smoking tobacco
* Using alcohol
* Having any chronic disease
* Having end-stage chronic renal failure
* Receiving chemotherapy and/or radiotherapy
* Being in menopausal, pregnant and/or lactation period,
* Using antioxidant vitamin and mineral supplements
* Following any diet program

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants who applied to Ankara City Hospital Endochronology Polyclinic between January and April 2021.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Serum native thiol level | Baseline (preprandial in the morning)
  serum native thiol level in μmol/L
Serum disulphide level | Baseline (preprandial in the morning)
  serum disulphide level in μmol/L
Serum total thiol level | Baseline (preprandial in the morning)
  serum total thiol level in μmol/L
Disulphide/native thiol ratio | Baseline (preprandial in the morning)
  Disulphide/native thiol ratio X (100 )
Disulphide/total thiol ratio | Baseline (preprandial in the morning)
  Disulphide/total thiol ratio X (100 )
Native thiol/total thiol ratio | Baseline (preprandial in the morning)
  Native thiol/total thiol ratio X (100 )
Dietary antioxidant capacity | Baseline
  Dietary intake assessed using 3-day dietary records. Participants instructed to record all dietary intake for 3 consecutive days, including 2 weekdays and 1 weekend day. Average value of 3 day nutrients were recorded and analyzed using Nutrition Data Base Ebispro for Windows, Stuttgart, Germany; Turkish Version (BeBiS 8.2), for Research software.

SECONDARY OUTCOMES:
Ischemia-modified albumin | Baseline (preprandial in the morning)
  ischaemia-modified albumin in ABSU
Dietary antioxidant intake | Baseline
  Dietary intake assessed using 3-day dietary records. Participants instructed to record all dietary intake for 3 consecutive days, including 2 weekdays and 1 weekend day. Average value of 3 day nutrients were recorded and analyzed using Nutrition Data Base Ebispro for Windows, Stuttgart, Germany; Turkish Version (BeBiS 8.2), for Research software.
Oxidative balance score | Baseline
  Dietary intake assessed using 3-day dietary records. Participants instructed to record all dietary intake for 3 consecutive days, including 2 weekdays and 1 weekend day. Average value of 3 day nutrients were recorded and analyzed using Nutrition Data Base Ebispro for Windows, Stuttgart, Germany; Turkish Version (BeBiS 8.2), for Research software.
Fasting plasma glucose | Baseline (preprandial in the morning)
  Fasting plasma glucose in mg/dL
hemoglobin A1c (HbA1c) | Baseline (preprandial in the morning)
  hemoglobin A1c (HbA1c) in %
Total cholesterol | Baseline (preprandial in the morning)
  Total cholesterol in mg/dL
Low-density lipoprotein (LDL) cholesterol | Baseline (preprandial in the morning)
  Low-density lipoprotein (LDL) cholesterol in mg/dL
High-density lipoprotein (HDL) cholesterol | Baseline (preprandial in the morning)
  High-density lipoprotein (HDL) cholesterol in mg/dL
Very low-density lipoprotein (VLDL) cholesterol | Baseline (preprandial in the morning)
  Very low-density lipoprotein (VLDL) cholesterol in mg/dL
non high-density lipoprotein (HDL) cholesterol | Baseline (preprandial in the morning)
  non high-density lipoprotein (HDL) cholesterol in mg/dL
total/high-density lipoprotein (HDL) cholesterol | Baseline (preprandial in the morning)
  total/high-density lipoprotein (HDL) cholesterol ratio
Triglyceride | Baseline (preprandial in the morning)
  Triglyceride in mg/dL
C-reactive protein | Baseline (preprandial in the morning)
  C-reactive protein in mg/dL
Body weight | Baseline
  Body weight in kg
Height | Baseline
  Height in meters
Body mass index | Baseline
  Body weight was measured via bioelectrical impedance analysis. Body height was taken by trained researcher in Frankfort Plane via Stadiometer. Weight and height combined to report body mass index in kg/m^2.
Fat mass | Baseline
  Fat mass in kg
Fat mass percentage | Baseline
  Fat mass percentage in %
Fat free mass | Baseline
  Fat free mass in kg
Total body water | Baseline
  Total body water in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No